CLINICAL TRIAL: NCT05492812
Title: Evaluation of the Effect of Chloral Hydrate, Hydroxyzine and Melatonin Used as Sedative Drugs in EEG Recording in Children
Brief Title: Sedation and Nursing Management in EEG Recording in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Serife Tutar, Assistant professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021
Record Dates: First submitted 2022-07-15; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Electroencephalography; Melatonin; Chloral Hydrate; Hydroxyzine; Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Chloral Hydrate; Hydroxyzine; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chloral Hydrate (Experimental): Chloral hydrate was administered orally to children at a dose of 25-50 mg/kg/dose. After the sedative drug administration, the child was taken to a quiet and dark sleep room in the polyclinic environment with his parents in order to enable the child to fall asleep. In this process, the child was evaluated by the nurse every 5 minutes with the Ramsay Sedation Score. Children with a Ramsay Sedation Score of 4-6 were taken to the EEG room for recording. During the sedation, the child's blood pressure, oxygen saturation and pulse were checked every 5 minutes. EEG electrodes were placed in accordance with the international 10-20 electrode positioning system. An average of 30 minutes of EEG recording was made for each patient. The awakening process of children whose EEG recordings were completed was evaluated with the Steward Recovery Score. Individuals with a score of 6 were accepted as awake, and the child's procedure was completed.
  Interventions: Other: Sedation and Nursing Management in EEG Recording in Children; Drug: Chloral Hydrate
- Hydroxyzine (Experimental): Hydroxyzine was administered orally to children at a dose of 1-2 mg/kg/dose. After the sedative drug administration, the child was taken to a quiet and dark sleep room in the polyclinic environment with his parents in order to enable the child to fall asleep. In this process, the child was evaluated by the nurse every 5 minutes with the Ramsay Sedation Score. Children with a Ramsay Sedation Score of 4-6 were taken to the EEG room for recording. During the sedation, the child's blood pressure, oxygen saturation and pulse were checked every 5 minutes. EEG electrodes were placed in accordance with the international 10-20 electrode positioning system. An average of 30 minutes of EEG recording was made for each patient. The awakening process of children whose EEG recordings were completed was evaluated with the Steward Recovery Score. Individuals with a score of 6 were accepted as awake, and the child's procedure was completed.
  Interventions: Other: Sedation and Nursing Management in EEG Recording in Children; Drug: Hydroxyzine
- Melatonin (Experimental): Melatonin was administered orally 3 mg up to 15 kilograms, and 6 mg after 15 kilograms.After the sedative drug administration, the child was taken to a quiet and dark sleep room in the polyclinic environment with his parents in order to enable the child to fall asleep. In this process, the child was evaluated by the nurse every 5 minutes with the Ramsay Sedation Score. Children with a Ramsay Sedation Score of 4-6 were taken to the EEG room for recording. During the sedation, the child's blood pressure, oxygen saturation and pulse were checked every 5 minutes. EEG electrodes were placed in accordance with the international 10-20 electrode positioning system. An average of 30 minutes of EEG recording was made for each patient. The awakening process of children whose EEG recordings were completed was evaluated with the Steward Recovery Score. Individuals with a score of 6 were accepted as awake, and the child's procedure was completed.
  Interventions: Other: Sedation and Nursing Management in EEG Recording in Children; Drug: Melatonin

INTERVENTIONS:
Other: Sedation and Nursing Management in EEG Recording in Children — Evaluation of the effect of sedative agents applied during EEG recording in children
Drug: Chloral Hydrate — Chloral Hydrate
  Arms: Chloral Hydrate
Drug: Hydroxyzine — Hydroxyzine
  Arms: Hydroxyzine
Drug: Melatonin — Melatonin
  Arms: Melatonin

SUMMARY:
Electroencephalogram (EEG) has an important place in establishing the correct diagnosis, providing appropriate intervention, and predicting the prognosis in the long term in children. When the literature is examined, it is seen that different sedative drugs (benzodiazepines, barbiturates, phenothiazine, chloral hydrate, hydroxyzine, melatonin, etc.) and their combinations are used to provide sedation during EEG recordings, but there is no ideal sedative drug. Nurses working in the field of pediatric neurology in EEG recordings; It has important roles in preparing the child and parent for the procedure, applying sedation before the procedure, performing the EEG recording properly, monitoring vital signs during the procedure, monitoring the effects of the sedative substance after the procedure, and sending the patient home safely. Pediatric nurses fulfill these roles by adopting a multidisciplinary team approach. In this context, the aim of our research is; The aim of this study is to evaluate the effects of chloral hydrate, hydroxyzine and melatonin, which are used as sedative agents before EEG recording in children, on sleep success, time to fall asleep, side effects and EEG background.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of chloral hydrate, hydroxyzine and melatonin, which are used as sedative agents before EEG recording in children, on sleep success, time to fall asleep, side effects and EEG background.It is a randomized controlled experimental study.The universe of the study consisted of all children who had EEG recordings in the Pediatric Neurology Outpatient Clinic of a tertiary hospital. Its sample is; It comprised 180 children aged 1-7 years who met the inclusion criteria, evaluated for epilepsy, suspected epilepsy, febrile convulsions, and other neurological diseases.G power program was used to determine the sample size of the study. For each group (chloral hydrate, hydroxyzine, melatonin and natural sleep) 45 individuals were included in the study by taking 95% power and 0.05 margin of error while making the calculation. Randomization was carried out in the study in order to provide an equal number of samples for each group (chloral hydrate, hydroxyzine, melatonin and natural sleep) and to avoid bias. "Block randomization method" was used in order to provide equal samples for all four groups in randomization.Data Collection tools of the research; Child's Information Form, Ramsay Sedation Score, Steward Recovery Score. Statistical analyzes of the study were performed with the SPSS 20.0 (IBM Incorp, Chicago, IL, USA) program. Descriptive measures were frequency (percentage ratio) for categorical variables, mean±SD and median for numerical variables; It was presented as Q1-Q3. Conformity of continuous numerical measurements to normal distribution was tested by Kolmogorov-Smirnov method, but it was found that it did not fit normal distribution (p <0.05). Multivariate logistic regression model was established to determine the properties that are effective on sedative substances. A p value of <0.05 was considered statistically significant in the entire study. In order to conduct the study, ethical approval from the Antalya Training and Research Hospital Clinical Research Ethics Committee, approval from the Turkish Medicines and Medical Devices Agency, institutional permission from the hospital where the study will be conducted, and written consent from the participants were obtained.

ELIGIBILITY:
Inclusion Criteria:

* According to the classification determined by the American Society of Anesthesiologist (ASA) (Dripps, 1963; Daabis, 2011), in the risk group of ASA I (normal healthy individual), ASA II (with mild systemic disease), the procedure preparation given by the EEG nurse is in accordance with the educational steps. The children who came to the shooting were included in the study.

Exclusion Criteria:

* Severe systemic disease (neurological, cardiac, respiratory, metabolic and gastrointestinal system), known hypersensitivity to the sedative agent, vomiting after sedative drug administration, waking up during the shooting, failing to fall asleep, and the procedure preparation training steps given by the EEG nurse Children who were not prepared properly were not included in the study.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Success in falling asleep | 12 month
  After the sedative drug administration, the child was taken to a quiet and dark sleep room in the polyclinic environment with his parents in order to enable the child to fall asleep. In this process, the child was evaluated by the nurse every 5 minutes with the Ramsay Sedation Score. Children with a Ramsay Sedation Score of 4-6 were taken to the electroencephalogram room for recording.
Sleep Time | 12 month
  After the sedative drug administration, the child was taken to a quiet and dark sleep room in the polyclinic environment with his parents in order to enable the child to fall asleep. In this process, the child was evaluated by the nurse every 5 minutes with the Ramsay Sedation Score. Children with a Ramsay Sedation Score of 4-6 were taken to the electroencephalogram room for recording.The time elapsed during this period was recorded as the time to fall asleep.
Ramsay Sedation Score on electroencephalogram background | 12 month
  After the sedative drug administration, the child was taken to a quiet and dark sleep room in the polyclinic environment with his parents in order to enable the child to fall asleep. In this process, the child was evaluated with the Ramsay Sedation Score. Children with a Ramsay Sedation Score of 4-6 were taken to the electroencephalogram room for recording. Electroencephalogram electrodes were placed in accordance with the international 10-20 electrode positioning system. An average of 30 minutes of electroencephalogram recording was made for each patient. Post-extraction records were evaluated by a pediatric neurologist and recorded in the data collection form.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Tutar, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will be shared after the research is published